CLINICAL TRIAL: NCT02058212
Title: Does Antioxidant Supplementation to Endometriotic Women Undergoing ICSI Could Alter Reactive Oxygen Species (ROS) Levels and Affect Pregnancy Outcome
Brief Title: Use of Antioxidant in Endometriotic Women to Improve Intracytoplasmic Sperm Injection (ICSI)
Acronym: ROS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, olfat nouh riad, assisstant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: antioxidants for endometriosis
Record Dates: First submitted 2014-02-05; First posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Endometriosis
Keywords: ICSI; antioxidants; ROS; endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Zinc; Selenium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no antioxidant , ROS , pregnancy outcome (Placebo Comparator): no anti oxidant in the form of ascorbate 1000mg, vitamin E 400, zinc and selenium) will be given to endometriotic women undergoing IVF
  Interventions: Drug: ascorbate 1000mg, vitamin E 400, zinc and selenium
- antioxidant , ROS , pregnancy outcome (Active Comparator): anti oxidant in the form of ascorbate 1000mg, vitamin E 400, zinc and selenium)
  Interventions: Drug: ascorbate 1000mg, vitamin E 400, zinc and selenium

INTERVENTIONS:
Drug: ascorbate 1000mg, vitamin E 400, zinc and selenium — anti oxidant in the form of ascorbate 1000mg, vitamin E 400, zinc and selenium) are given to half patients only before IVF , plasma level of ROS are detected before and on day of oocyte retrieval then correlated to pregnancy outcome

SUMMARY:
ROS plays an essential role in the pathogenesis of many reproductive processes. High follicular fluid ROS levels are associated with negative IVF outcomes.

is plasma level of reactive oxygen species is affected by antioxidant treatment in endometriotic women?

DETAILED DESCRIPTION:
Study design, size, duration: : prospective randomized controlled clinical trial 50 patients with endometriosis diagnosed by US prepared for ICSI were enrolled in the study after consent. they were randomized into 2 groups 25 received antioxidants before starting the protocol , 25 did not receive . randomization was done by closed envelop single blind for patient Participants/materials, setting, methods: was done in the Egyptian centre for IVF from March 2013 to October 2013 . 50 patients with endometriosis diagnosed by US prepared for ICSI were enrolled in the study after consent. they were randomized into 2 groups 25 received antioxidants before starting the protocol , 25 did not receive . all patients were subjected to plasma sample before start long protocol for induction and second on day of ovum pick up . embryo transfer was done according to embryo grading .

ELIGIBILITY:
Inclusion Criteria:

* patients with endometriosis

Exclusion Criteria:

patients with no endometriosis , not suitable for ICSI-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
plasma reactive oxygen species affection by antioxidant treatment | 3 months
  measure before and 3months after antioxidant treatment

SECONDARY OUTCOMES:
clinical pregnancy rate | 2 months
  long protocol administration

CONTACTS AND LOCATIONS:
Overall Officials: olfat nouh riad, MD, Principal Investigator
Locations (2):
- Egypt (2):
  - egyption centre for IVF, Maadi
  - Maadi